CLINICAL TRIAL: NCT00315445
Title: A Comparative Study of Buprenorphine TDS, Oxycodone/ Acetaminophen Tablets Qid and Placebo in Patients With Chronic Back Pain
Brief Title: The Safety and Efficacy of the Buprenorphine Transdermal System (BTDS) in Subjects With Chronic Back Pain.
Acronym: BP96-0604
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Medical Director, Medical Research, Purdue Pharma L.P.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP96-0604
Record Dates: First submitted 2006-04-17; First posted 2006-04-18 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Back Pain
Keywords: chronic back pain; opioid; transdermal
MeSH Terms: conditions — Back Pain | interventions — Buprenorphine; Acetaminophen; tyramine-deoxysorbitol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Placebo oxycodone (OXY)/acetaminophen (APAP) tablets and placebo transdermal patch (TDS) 5, 10, or 20
  Interventions: Drug: Placebo oxycodone/acetaminophen tablets; Drug: Placebo transdermal patch (TDS)
- OXY/APAP (Active Comparator): 5 mg oxycodone/325 mg acetaminophen tablets
  Interventions: Drug: OXY/APAP
- BTDS (Experimental): Buprenorphine transdermal patch 5, 10, or 20 mcg/hour
  Interventions: Drug: Buprenorphine transdermal patch

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine 5, 10, or 20 mcg/hour patch applied transdermally for 7-day wear.
  Other Names: Butrans™
  Arms: BTDS
Drug: Placebo oxycodone/acetaminophen tablets — Placebo oxycodone/acetaminophen tablets; 1, 2, or 3 tablets taken four times/day.
  Arms: Placebo
Drug: OXY/APAP — 5 mg oxycodone / 325 mg acetaminophen tablets; 1, 2, or 3 tablets taken four times/day.
  Arms: OXY/APAP
Drug: Placebo transdermal patch (TDS) — Placebo transdermal patch 5, 10, or 20 applied transdermally for 7-day wear
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the safety of the buprenorphine transdermal system (5, 10, and 20) in comparison to placebo transdermal system and immediate release oxycodone/ acetaminophen in subjects with chronic back pain. The double-blind treatment intervention duration is 84 days during which time supplemental analgesic medication (non-steroidal anti-inflammatory drugs) will be allowed for all subjects in addition to study drug.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over twenty-five years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* clinical evidence of stable, chronic (>2 months) back pain related to intervertebral disc disease, nerve root entrapment, spondylolithesis, and osteoarthritis or other, similar nonmalignant conditions.
* unacceptable pain control despite currently taking a nonsteroidal anti-inflammatory drug considered at a therapeutic and/or tolerated dose or, subjects currently taking </=2 short-acting opioid doses per day, or subjects taking 3-12 short-acting opioid doses per day.

Exclusion Criteria:

* receiving opioids at an average daily dose of >90 mg of oral morphine equivalents or receiving more than 12 tablets per day of short-acting opioid-containing products.
* scheduled to have surgery (including dental) involving the use of preoperative or postoperative analgesics or anesthetics during the study period.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 1997-12; Primary Completion 1998-05 (Actual); Study Completion 1998-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Phoenix Center for Clinical Research, Phoenix, Arizona
  - Phoenix Orthopedic Center, Ltd., Phoenix, Arizona
  - Gainesville Clinical Research Center, Gainesville, Florida
  - SeaView Research, Miami, Florida
  - Park Place Therapeutic Center, Plantation, Florida
  - Atlanta Research Center, Decatur, Georgia
  - The Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - New Jersey Research Foundation, Linwood, New Jersey
  - North Carolina Clinical Research, Inc., Raleigh, North Carolina
  - Research Across America, Dallas, Texas
  - Metroplex Clinical Research Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10-Dec-1997 (first subject, first visit) to 08-May-1998 (last subject last visit) in 13 centers in the United States
Pre-assignment Details: This study was designed to evaluate the efficacy and safety of BTDS in comparison with current pharmacotherapeutic pain management practice and placebo in opioid-naïve or opioid-experienced adult subjects with chronic back pain not manageable with nonopioid analgesics alone (range, 19-85 years).
Groups:
- Placebo: Placebo oxycodone/acetaminophen (APAP) 1, 2, or 3 tablets four times/day and transdermal patch (TDS) placebo 5, 10, or 20 applied for 7-day wear.
- OXY/APAP: 5 mg oxycodone/325 mg acetaminophen, 1, 2, or 3 tablets four times/day.
- BTDS: Buprenorphine transdermal patch 5, 10, or 20 mcg/hour applied for 7-day wear.
Period: Overall Study
Arm/Group | Placebo | OXY/APAP | BTDS
Started | 45 | 43 | 46
Completed | 18 | 27 | 22
Not Completed | 27 | 16 | 24
Not completed — Adverse Event | 7 | 12 | 15
Not completed — Lack of Efficacy | 16 | 1 | 7
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 1
Not completed — Other | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | OXY/APAP | BTDS | Total
Number analyzed (Participants) | 45 | 43 | 46 | 134
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (2.2) | 49 (2.5) | 54 (2.2) | 52 (1.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 28 | 80
  Male | 20 | 16 | 18 | 54
Opioid Experience [Number; unit: participants] — Subjects were either classified as "opioid naive" (those not currently receiving an opioid-containing analgesic or those receiving 2 or fewer short-acting opioid tablets or capsules per day) or "opioid experienced" (those receiving a controlled-release opioid analgesic at a dose of ≤ 90 mg of morphine equivalents per day or those receiving 3 to 12 capsules or tablets of short-acting opioid analgesics per day)
  participants
    Opioid naive | 39 | 34 | 34 | 107
    Opioid experienced | 6 | 9 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Pain on the Average, Mean Change From Baseline Days 21-84 (Last Observation Carried Forward [LOCF])
Description: Subjects were asked, "Please rate your pain by circling the one number (0-10) that best describes your pain on the average since your last visit." 0 = no pain and 10 = pain as bad as you can imagine it.
Time Frame: On baseline day 1 and days 21, 30, 45, 60, 75, and 84, and, if applicable, at early termination.
Population: All 134 subjects randomized and received study drug were included in the intent-to-treat (ITT) and safety analyses. ITT Subjects With Efficacy Data (N = 133) 1 subject was withdrawn from study because the informed consent was never obtained. This subject had no efficacy data but was included the analysis of discontinuation due to lack of efficacy.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | -1.01 (0.37) | -1.82 (0.36) | -1.92 (0.34)
Statistical Analysis 1: Comparison: Placebo vs BTDS; A repeated measures analysis was performed to assess the effects due to treatment, center, and treatment by center interaction. Observations within each subject were assumed to follow a first-order autoregressive model. Missing values were extrapolated by the last observation carried forward (LOCF). Covariates were gender, age, race, weight, baseline pain, and previous opioid use which were incorporated into the model when P < 0.10, using a backward elimination procedure; Test type: Superiority or Other; p = 0.0350, Mixed Models Analysis — P values are from a repeated measures model
Statistical Analysis 2: Comparison: Placebo vs OXY/APAP; Test type: Superiority or Other; p = 0.0624, Mixed Models Analysis — Repeated measures analysis to assess the effects due to treatment, center, and treatment by center. Missing values = last observation carried forward (LOCF). Covariates: gender, age, race, weight, baseline pain, and previous opioid use

2. Secondary Outcome: "Physical Functioning" Scale of the Medical Outcomes Survey (MOS) 36 Item Short-Form Health Survey (SF-36): Mean Percent ± Standard Error of the Mean (SEM) at Day 84 (LOCF)
Description: The Medical Outcomes Survey (MOS) Short-Form-36 Health Survey (SF-36) assesses 8 categories of functionality through 36 individual questions. "Physical Functioning" is 1 of the 8 categories. Its transformed score, scaled from 0% to 100%, is used. A higher score represents a better subject condition. The survey was completed by the subject at the clinic. The mean scores were analyzed.
Time Frame: Day 84, or, if applicable, at early termination
Population: All 134 subjects who were randomized and received study drug were included in the intent-to-treat and safety analyses. No subjects were excluded.
  Intent-to-treat Subjects With Efficacy Data (N = 133) 1 subject was withdrawn from the study because the informed consent was never obtained.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | 46.4 (4.0) | 44.5 (3.9) | 46.5 (3.6)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 46.4, 90% CI 2-sided [40.2 to 48.7]
Statistical Analysis 2: Comparison: OXY/APAP; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 44.5, 90% CI 2-sided [43.3 to 52.4]
Statistical Analysis 3: Comparison: BTDS; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 46.5, 90% CI 2-sided [41.7 to 50.2]

3. Secondary Outcome: "Physical Role" Scale (MOS SF-36): Mean Percent ± SEM at Day 84(LOCF)
Description: The Medical Outcomes Survey Short-Form-36 health survey assesses 8 categories of functionality through 36 individual questions. "Physical Role" is 1 of the 8 categories. Its transformed score, scaled from 0% to 100%, is used. A higher score represents a better subject condition. The survey was completed by the subject at the clinic. The mean scores were analyzed.
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | 18.9 (4.8) | 24.4 (5.9) | 33.9 (5.8)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 18.9, 90% CI 2-sided [5.2 to 26.2]
Statistical Analysis 2: Comparison: OXY/APAP; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 24.4, 90% CI 2-sided [10.7 to 32.0]
Statistical Analysis 3: Comparison: BTDS; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 33.9, 90% CI 2-sided [16.0 to 35.2]

4. Primary Outcome: Pain Right Now, Mean Change From Baseline, Days 21-84 (LOCF)
Description: Subjects were asked, "Please rate your pain by circling the one number (0-10) that tells how much pain you have right now." Subjects rated their answers on a 0-10 ordinal scale from 0 = "No pain" to 10 = "Pain as bad as you can imagine it." Pain right now is presented as the LSmean [change from baseline] (SE).
Time Frame: Assessed at baseline day 1 and days 21, 30, 45, 60, 75, and 84, and, if applicable, at early termination.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | -0.80 (0.38) | -1.53 (0.37) | -1.66 (0.34)
Statistical Analysis 1: Comparison: Placebo vs BTDS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0452, Mixed Models Analysis — Multiple linear regression
Statistical Analysis 2: Comparison: Placebo vs OXY/APAP; Test type: Superiority or Other; p = 0.0962, Mixed Models Analysis

5. Secondary Outcome: "Bodily Pain" (MOS SF-36): Mean Percent at Day 84 (LOCF)
Description: The MOS Short-Form Health Survey assesses 8 categories of functionality through 36 individual questions. "Bodily Pain" is 1 of the 8 categories. Its transformed score, scaled from 0% to 100%, is used. A higher score represents a better subject condition. The survey was completed by the subject at the clinic. The mean scores were analyzed.
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | 35.3 (3.1) | 39.0 (3.4) | 41.9 (3.1)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 35.3, 90% CI 2-sided [24.3 to 35.6]
Statistical Analysis 2: Comparison: OXY/APAP; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 39.0, 90% CI 2-sided [29.0 to 40.3]
Statistical Analysis 3: Comparison: BTDS; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 41.9, 90% CI 2-sided [32.1 to 42.5]

6. Secondary Outcome: "General Health" (MOS SF-36): Mean Percent ± SEM at Day 84 (LOCF)
Description: The MOS Short-Form Health Survey assesses 8 categories of functionality through 36 individual questions. "General Health" is 1 of the 8 categories. Its transformed score, scaled from 0% to 100%, is used. A higher score represents a better subject condition. The survey was completed by the subject at clinic. The mean scores were analyzed.
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | 52.4 (3.5) | 52.5 (3.5) | 57.7 (3.4)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 52.4, 90% CI [50.3 to 56.6]
Statistical Analysis 2: Comparison: OXY/APAP; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 52.5, 90% CI 2-sided [51.8 to 58.3]
Statistical Analysis 3: Comparison: BTDS; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 57.7, 90% CI 2-sided [52.3 to 58.6]

7. Secondary Outcome: "Vitality" (MOS SF-36): Mean Percent ± SEM at Day 84 (LOCF)
Description: The MOS Short-Form Health Survey assesses 8 categories of functionality through 36 individual questions. "Vitality" is 1 of the 8 categories. Its transformed score, scaled from 0% to 100%, is used. A higher score represents a better subject condition. The survey was completed by the subject at the clinic. The mean scores were analyzed.
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | 39.0 (3.7) | 42.9 (3.7) | 41.2 (3.5)

8. Secondary Outcome: "Social Functioning" (MOS SF-36): Mean Percent ± SEM at Day 84 (LOCF)
Description: The MOS Short-Form Health Survey assesses 8 categories of functionality through 36 individual questions. "Social Functioning" is 1 of the 8 categories. Its transformed score, scaled from 0% to 100%, is used. A higher score represents a better subject condition. The survey was completed by the subject at the clinic.
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | 53.3 (4.2) | 59.5 (3.9) | 65.2 (4.4)

9. Secondary Outcome: "Emotional Role" (MOS SF-36): Mean Percent ± SEM at Day 84 (LOCF)
Description: The MOS Short-Form Health Survey assesses 8 categories of functionality through 36 individual questions. "Emotional Role" is 1 of the 8 categories. Its transformed score, scaled from 0% to 100%, is used. A higher score represents a better subject condition. The survey was completed by the subject at the clinic.
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | 55.3 (6.7) | 56.3 (7.1) | 63.0 (6.2)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 55.3, 90% CI 2-sided [49.8 to 67.9]
Statistical Analysis 2: Comparison: OXY/APAP; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 56.3, 90% CI 2-sided [45.9 to 65.3]
Statistical Analysis 3: Comparison: BTDS; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 63.0, 90% CI 2-sided [53.1 to 70.9]

10. Secondary Outcome: "Mental Health" (MOS SF-36):Mean Percent ± SEM at Day 84 (LOCF)
Description: The MOS Short-Form Health Survey assesses 8 categories of functionality through 36 individual questions. "Mental Health" is 1 of the 8 categories. Its transformed score, scaled from 0% to 100%, is used. A higher score represents a better subject condition. The survey was completed by the subject at the clinic.
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | 67.4 (3.1) | 68.8 (2.7) | 67.8 (3.3)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 67.4, 90% CI 2-sided [61.3 to 68.6]
Statistical Analysis 2: Comparison: OXY/APAP; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 68.8, 90% CI 2-sided [61.7 to 68.8]
Statistical Analysis 3: Comparison: BTDS; Test type: Superiority or Other; Day 84 Mean; Day 84 Mean = 67.8, 90% CI 2-sided [62.0 to 68.7]

11. Secondary Outcome: Therapeutic Response - Investigator: Mean ± SEM (Day 84)(LOCF)
Description: The therapeutic response was rated by the investigator. The assessment was completed by the investigator using a 0-3 ordinal scale from 0 = "No response" to 3 = "Marked response."
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 35 | 34 | 34
Units on a scale | 1.1 (0.2) | 2.0 (0.2) | 1.9 (0.2)

12. Secondary Outcome: Therapeutic Response - Subject: Mean ± SEM (Day 84) (LOCF)
Description: The therapeutic response was rated by the subject. The assessment was completed by the subject using a 0-3 ordinal scale from 0 = "No response" to 3 = "Marked response."
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 36 | 34 | 33
Units on a scale | 1.1 (0.2) | 2.1 (0.1) | 2.0 (0.2)

13. Secondary Outcome: Subject Comparison to Prestudy Analgesic: Mean ± SEM (Day 84)(LOCF)
Description: The subject compared study drug treatment to prestudy analgesic. The assessment was completed by the subject using a 0-2 ordinal scale from 0 = "Worse than prestudy medicine" to 2 = "Better than prestudy medicine."
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 36 | 34 | 33
Units on a scale | 0.9 (0.1) | 1.4 (0.1) | 1.4 (0.1)

14. Secondary Outcome: Subject Satisfaction: Mean ± SEM (Day 84)(LOCF)
Description: The subject assessed satisfaction with study drug. The assessment was completed by the subject using a 0-3 ordinal scale from 0 = "No response" to 3 = "Marked response."
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 36 | 34 | 33
Units on a scale | 2.2 (0.1) | 1.8 (0.1) | 1.7 (0.2)

15. Secondary Outcome: Time to Stable Pain Management
Description: For each subject, "time to stable pain management" is defined as the first (post-baseline) time during the titration period when his/her "diary pain" was 4 or less (or at least 2 points lower than baseline) for 3 consecutive daily records or the "pain on the average" (at the day 7 or day 21 visit) was 4 or less (or at least 2 points lower than baseline).
Time Frame: Start of study to day 21.
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Days | 14 [4 to NA] — NA because less than 75% of placebo subjects achieved stable pain management. | 7 [4 to 13] | 7 [4 to 18]
Statistical Analysis 1: Comparison: Placebo vs BTDS; Test type: Superiority or Other; p = 0.054, Regression, Cox; For the secondary outcome measure no alpha adjustment for multiple comparison was performed; Hazard Ratio (HR) = 1.67
Statistical Analysis 2: Comparison: Placebo vs OXY/APAP; Test type: Superiority or Other; p = 0.138, Regression, Cox; For the secondary outcome measure no alpha adjustment for multiple comparison was performed; Hazard Ratio (HR) = 1.51

16. Secondary Outcome: The Time to Discontinuation Due to Lack of Efficacy
Description: Dropouts due to various reasons were summarized by counts and percentage. Cox proportional hazards regression was used to assess the treatment differences in time to dropout due to lack of efficacy. Clinically important covariates (including gender, age, race, weight, baseline pain, and previous opioid use) were incorporated into the model when statistically significant at P< .10, using a backward elimination procedure.
Time Frame: Time after dosing to dropout due to lack of efficacy
Population: All 134 subjects who were randomized and received study drug were included in the intent-to-treat and safety analyses. No subjects were excluded.
  Intent-to-treat Subjects With Efficacy Data (N = 133) 1 subject was withdrawn because the informed consent was never obtained and had no efficacy data.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Days | NA [21 to NA] — NA because few subjects (16 in the placebo group) experienced lack of efficacy during the study. | NA [NA to NA] — NA because few subjects (1 in the OXY/APAP group) experienced lack of efficacy during the study. | NA [NA to NA] — NA because few subjects (7 in the BTDS group) experienced lack of efficacy during the study.
Statistical Analysis 1: Comparison: Placebo vs BTDS; Test type: Superiority or Other; p = 0.0105, Regression, Cox; For the secondary outcomes no alpha adjustment for multiple comparison was performed; Hazard Ratio (HR) = 0.30
Statistical Analysis 2: Comparison: Placebo vs OXY/APAP; Test type: Superiority or Other; p = 0.0024, Regression, Cox; For the secondary outcome measure no alpha adjustment for multiple comparison was performed; Hazard Ratio (HR) = 0.04

17. Post Hoc Outcome: Sensitivity Analysis: "Pain on the Average" Change From Baseline in the Maintenance Period (Days 21 - 84) Baseline Observation Carried Forward (BOCF)
Description: as for outcome 1
Time Frame: Baseline to days 21 - 84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | -0.77 (0.38) | -1.70 (0.38) | -1.74 (0.35)
Statistical Analysis 1: Comparison: Placebo vs BTDS; Test type: Superiority or Other; p = .033, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs OXY/APAP; Test type: Superiority or Other; p = .043, Mixed Models Analysis

18. Post Hoc Outcome: Sensitivity Analysis: "Pain Right Now" Change From Baseline in the Maintenance Period (Days 21-84), BOCF
Description: Subjects were asked, "Please rate your pain by circling the one number (0-10) that tells how much pain you have right now." Subjects rated their answers on a 0-10 ordinal scale from 0 = "No pain" to 10 = "Pain as bad as you can imagine it." Primary back pain was measured.
Time Frame: Baseline to days 21-84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | -0.53 (0.37) | -1.46 (0.37) | -1.64 (0.33)
Statistical Analysis 1: Comparison: Placebo vs BTDS; Test type: Superiority or Other; p = .011, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs OXY/APAP; Test type: Superiority or Other; p = .034, Mixed Models Analysis

19. Post Hoc Outcome: Sensitivity Analysis "Pain on the Average" Change From Baseline in the Maintenance Period (Days 21-84) (Hybrid BOCF/LOCF)
Description: Subjects were asked, "Please rate your pain by circling the one number (0-10) that best describes your pain on the average since your last visit." 0 = no pain and 10 = pain as bad as you can imagine it.
  This is a multiple imputation method that requires imputed changes from baseline to be stratified by discontinuation (D/C) reason. If subject D/C'd due to AE, the baseline observation was carried forward (ie, BOCF method of imputation). If subject D/C'd other than for an AE, the last missing data prior to D/C of study drug was carried forward (ie, LOCF method of imputation).
Time Frame: Baseline to days 21-84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | -0.91 (0.39) | -1.77 (0.39) | -1.86 (0.35)
Statistical Analysis 1: Comparison: Placebo vs BTDS; Test type: Superiority or Other; p = .038, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs OXY/APAP; Test type: Superiority or Other; p = 0.63, Mixed Models Analysis

20. Post Hoc Outcome: Sensitivity Analysis: "Pain Right Now" Change From Baseline in the Maintenance Period (Days 21-84) (Hybrid BOCF/LOCF)
Description: Subjects were asked, "Please rate your pain by circling the one number (0-10) that tells how much pain you have right now." Subjects rated their answers on a 0-10 ordinal scale from 0 = "No pain" to 10 = "Pain as bad as you can imagine it."
  This is a multiple imputation method that requires imputed changes from baseline to be stratified by discontinuation (D/C) reason. If subject D/C'd from study due to AE, the baseline observation was carried forward (BOCF). If subject D/C'd from study other than for AE, the last missing data prior to D/C of study drug was carried forward (LOCF).
Time Frame: Baseline to days 21-84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | -0.78 (0.38) | -1.60 (0.38) | -1.59 (0.34)
Statistical Analysis 1: Comparison: Placebo vs BTDS; Test type: Superiority or Other; p = .064, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs OXY/APAP; Test type: Superiority or Other; p = .066, Mixed Models Analysis

21. Post Hoc Outcome: Sensitivity Analysis: "Pain on the Average" Change From Baseline to End of Treatment (Day 84) (Hybrid BOCF/LOCF)
Description: as for outcome 19
Time Frame: Baseline to day 84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | -1.44 (0.44) | -1.47 (0.44) | -1.70 (0.40)
Statistical Analysis 1: Comparison: Placebo vs BTDS; Test type: Superiority or Other; p = .607, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs OXY/APAP; Test type: Superiority or Other; p = .940, Mixed Models Analysis

22. Post Hoc Outcome: Sensitivity Analysis: "Pain Right Now" Change From Baseline to End of Treatment (Day 84) (Hybrid BOCF/LOCF)
Description: as for outcome 20
Time Frame: Baseline to day 84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | OXY/APAP | BTDS
Number analyzed (Participants) | 45 | 42 | 46
Units on a scale | -1.30 (0.45) | -1.56 (0.45) | -1.50 (0.41)
Statistical Analysis 1: Comparison: Placebo vs BTDS; Test type: Superiority or Other; p = .702, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs OXY/APAP; Test type: Superiority or Other; p = .634, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were followed until resolved or etiology diagnosed. Deaths, adverse events and discontinuations occurring more than 7 days after discontinuation of study medication were reported.
Description: AEs were learned of by spontaneous reports, subject interview, and daily diary.
Arm/Group | Placebo | OXY/APAP | BTDS
Serious Adverse Events (participants affected / at risk) | 2/45 | 3/43 | 3/46
Other Adverse Events (participants affected / at risk) | 20/45 | 35/43 | 37/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | OXY/APAP (N=43) | BTDS (N=46)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fractured humerous (Investigations) | 0 (0) | 1 (1) | 0 (0)
Increased back pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructed right kidney (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=45) | OXY/APAP (N=43) | BTDS (N=46)
Asthenia (General disorders) | 1 | 3 | 2
Fever (General disorders) | 0 | 1 | 3
Headache (General disorders) | 6 | 7 | 13
Pain abdomen (General disorders) | 3 | 2 | 1
Pain back (General disorders) | 1 | 1 | 5
Constipation (Gastrointestinal disorders) | 7 | 14 | 10
Dry mouth (Gastrointestinal disorders) | 5 | 9 | 10
Dyspepsia (Gastrointestinal disorders) | 4 | 1 | 6
Nausea (Gastrointestinal disorders) | 6 | 19 | 17
Vomiting (Gastrointestinal disorders) | 0 | 12 | 12
Edema peripheral (Metabolism and nutrition disorders) | 1 | 1 | 3
Dizziness (Nervous system disorders) | 7 | 14 | 14
Insomnia (Nervous system disorders) | 2 | 4 | 1
Somnolence (Nervous system disorders) | 4 | 17 | 12
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Sweating (Skin and subcutaneous tissue disorders) | 1 | 4 | 4
Dysuria (Renal and urinary disorders) | 0 | 3 | 0
Accidental injury (General disorders) | 1 | 4 | 2
Pain (General disorders) | 1 | 0 | 4
Tremor (Nervous system disorders) | 0 | 1 | 3
Pruritus at site (Skin and subcutaneous tissue disorders) | 7 | 9 | 7
Rash at site (Skin and subcutaneous tissue disorders) | 2 | 3 | 2
Infection (Infections and infestations) | 2 | 7 | 2

LIMITATIONS AND CAVEATS:
There was a large percentage of discontinuations across treatment groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days